CLINICAL TRIAL: NCT00333905
Title: The Effect of Ischemic Training on Exercise Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F4096R
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2006-06

CONDITIONS: Heart Failure; Congestive Heart Failure; Cardiovascular Disease
Keywords: Exercise; Exercise Therapy
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Motor Activity

INTERVENTIONS:
Procedure: Ischemic exercise training

SUMMARY:
The purpose of this study is to determine if reducing blood flow to an exercising muscle during exercise training will enhance the training effect on that muscle in people who have limited exercise because of congestive heart failure

DETAILED DESCRIPTION:
The objective of this study is to determine whether reduction of blood flow during stair-stepping and cycling ergometer leg exercise will contribute to an improvement in whole body exercise capacity or submaximal exercise endurance in patients with mild congestive heart failure. Two groups of 25 patients with mild to moderate CHF, aged 30-70, will be trained for 12 weeks. The experimental group will train with pressure cuffs inflated on one thigh and lower leg during exercise. The cuff will be applied on alternate legs during training, such that each leg has the same duration of ischemic training. The control group will train for a similar duration and intensity without pressure cuffs on the legs. Pre and post training measures will include VO2peak, exercise duration at 30% VO2peak, 6 minute walk test, Minnesota Living with Heart Failure questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Mild Congestive Heart Failure
* Must be able to exercise

Exclusion Criteria:

* Venous or arterial thrombus
* Lower extremity arthritis
* Blood clotting abnormalities
* Claudication
* Peripheral vascular disease
* Evidence of deep vein thrombosis on ultrasound

Ages: 30 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-03; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Exercise duration before and after 12 weeks of training during a submaximal exercise test and distance walked on a 6-minute walk test.

SECONDARY OUTCOMES:
Peak cycle ergometer VO2max test before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Milton V Icenogle, MD, Principal Investigator — Cardiology Division Chief, Medicine Service VAMC Albuquerque (501) Albuquerque, NM
Locations (1):
- New Mexico VA Health Care System, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Loeppky JA, Gurney B, Kobayashi Y, Icenogle MV. Effects of ischemic training on leg exercise endurance. J Rehabil Res Dev. 2005 Jul-Aug;42(4):511-22. doi: 10.1682/jrrd.2004.06.0069. PMID 16320146